CLINICAL TRIAL: NCT02436954
Title: Impact of Neuromuscular Blockade on Cerebral Oxygen Saturation in Laparoscopic Surgery Employ Carbon Dioxide-pneumoperitoneum
Brief Title: Regional Cerebral Oxygen Saturation in Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUH1160084
Record Dates: First submitted 2015-03-18; First posted 2015-05-07 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Cholecyctitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO2 insufflation at intra-abdominal pressure 8 mmHg (Placebo Comparator): CO2 insufflation with intra-abdominal pressure 8 mmHg during deep-NMB
  Interventions: Procedure: CO2 insufflation at intra-abdominal pressure 8 mmHg
- CO2 insufflation at intra-abdominal pressure 12 mmHg (Active Comparator): CO2 insufflation with intra-abdominal pressure 12 mmHg during deep-NMB
  Interventions: Procedure: CO2 insufflation at intra-abdominal pressure 12 mmHg

INTERVENTIONS:
Procedure: CO2 insufflation at intra-abdominal pressure 8 mmHg — insufflation of CO2 gas into peritoneum for maintaining the pressure of 8 mmHg
  Arms: CO2 insufflation at intra-abdominal pressure 8 mmHg
Procedure: CO2 insufflation at intra-abdominal pressure 12 mmHg — insufflation of CO2 gas into peritoneum for maintaining the pressure of 12 mmHg
  Arms: CO2 insufflation at intra-abdominal pressure 12 mmHg

SUMMARY:
While few studies have determined the optimal intra-abdominal CO2 insufflation pressure to achieve optimal surgical condition during LCs with deep-NMB and moderate-NMB in laparoscopic cholecystectomy (LC), previous studies suggested that the use of deep neuromuscular blockade (deep-NMB) can improve surgical condition and reduce the pressure for CO2 insufflation to achieve "optimal surgical space condition".

this difference in the pressure of intra-abdominal CO2 insufflation due to different strategies employing deep-NMB and moderate-NMB for LC may produce possible difference in patient's respiratory pattern and cerebral oxygenation. Although previous study (studies) showed that intra-abdominal CO2 insufflation (10-12 mmHg) decreases cerebral oxy-hemoglobin (HbO2) and total Hb measured by near-infrared spectroscopy (NIRS) during laparoscopic cholecystectomy (LC), few studies have speculated possible impact of different degree of NMB and intra-abdominal CO2 insufflation pressure on patient's cardiorespiratory profile and cerebral oxygenation, so far.

The present study determines and compares the changes CO2 absorption and cerebral oxygenation (cerebral perfusion) after applying CO2 insufflation with different intra-peritoneal pressure 8 vs 12 mmHg during deep-NMB.

ELIGIBILITY:
Inclusion Criteria:

* cholecystitis
* provision of written informed consent

Exclusion Criteria:

* COPD
* asthma
* low LV ejection fraction

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
regional cerebral oxygen saturation 1 | 1 min
  1 min after the initiation of pneumoperitonium
regional cerebral oxygen saturation 2 | 2 min
  2 min after the initiation of pneumoperitonium
regional cerebral oxygen saturation 3 | 3 min
  2 min after the initiation of pneumoperitonium

SECONDARY OUTCOMES:
end-tidal carbon dioxide 1 | 1 min
end-tidal carbon dioxide 2 | 2 min
end-tidal carbon dioxide 3 | 3 min
repiratory rate | 3 min